CLINICAL TRIAL: NCT01012258
Title: Open-label, Single-arm, Multicenter, Phase III Trial to Assess the Antitumor Activity and Safety of Cetuximab When Given in Combination With Radiotherapy for the Treatment of Locally Advanced Squamous Cell Carcinoma of the Head and Neck in Chinese Subjects
Brief Title: Cetuximab With Radiotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck in Chinese Subjects
Acronym: CHANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR62241-054
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: antitumor activity; safety; cetuximab in combination with radiotherapy; locally advanced squamous cell head & neck carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental): All eligible subjects will receive cetuximab treatment only during week 1 of the treatment course and concomitant cetuximab and boost radiotherapy (RT) during week two to week seven of the treatment course
  Interventions: Biological: Cetuximab + concomitant boost radiotherapy

INTERVENTIONS:
Biological: Cetuximab + concomitant boost radiotherapy — Cetuximab 400 milligram/square meter (mg/m^2) intravenous (IV) infusion over 120 minutes for 1 week, subsequently followed by 250 mg/m^2 IV infusion over 60 minutes, from week 2 to 7 along with concomitant boost radiotherapy: 72.0 Gray (Gy) total for 42 fractions in 6 weeks, initially
  * Once-daily fractions: 32.4 Gy in 18 fractions of 1.8 Gy for 3.6 weeks (5 fractions/week), followed by
  * Twice-daily fractions 39.6 Gy in 24 fractions for 2.4 weeks: morning dose 1.8 Gy/fraction for a total of 12 fractions 5 fractions/week; evening dose 1.5 Gy/fraction for a total of 12 fractions 5 fractions/week. Doses are separated by at least a 6-hour interval
  Other Names: Erbitux®

SUMMARY:
Primary objective: to assess the antitumor activity and safety profile of cetuximab when given in combination with radiotherapy (RT) for the treatment of locally advanced squamous cell carcinoma of the head and neck (SCCHN) in Chinese subjects.

Secondary objective: to assess the pharmacokinetic (PK) profile and immunogenicity of cetuximab in Chinese subjects.

Further objective: to identify for cetuximab potential predictive biomarkers of response and safety.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient greater than or equal to (>=) 18 years of age
* Pathologically proven squamous cell carcinoma arising in the oropharynx, hypopharynx or larynx
* Stage III or IV disease with an expected survival of at least 12 months
* Medically suitable to withstand a course of concomitant boost RT
* Presence of at least 1 bi-dimensionally measurable lesion identified either by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to modified World Health Organization (WHO) criteria
* Karnofsky Performance Status (KPS) >=80 at trial entry
* Neutrophils >=1.5*10^9/Liter (L), platelet count >= 100*10^9/L, hemoglobin >= 90 gram/liter (g/L)
* Total bilirubin less than or equal to (<=) 2*upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3*ULN
* Serum creatinine <=133 micromole/liter (mcmol/L)
* Serum calcium within normal range
* Effective contraception if procreative potential exists (applicable to both male and female subjects)
* Chinese with Chinese citizenship
* Signed written informed consent

Exclusion Criteria:

* Evidence of distant metastatic disease
* Squamous cell carcinoma arising in the nasopharynx or oral cavity
* Receipt of prior systemic chemotherapy within the last 3 years
* Previous surgery for the tumor under study other than biopsy
* Receipt of prior RT to the head and neck
* Currently receiving RT as part of a postoperative regimen following primary surgical resection
* Planned neck dissection after trial RT
* Active infection (infection requiring IV antibiotics), including active tuberculosis, or known and declared human immunodeficiency virus (HIV)
* Uncontrolled diabetes mellitus, pulmonary fibrosis, acute pulmonary disorder, interstitial pneumonia, cardiac failure or liver failure
* Uncontrolled hypertension defined as systolic blood pressure >=180 millimeter of mercury (mmHg) and/or diastolic blood pressure >=130 mmHg under resting conditions
* Pregnancy (absence to be confirmed by serum beta human chorionic gonadotrophin [beta-HCG] test) or breastfeeding
* Concomitant chronic systemic immune therapy or hormonal therapy as cancer therapy
* Other concomitant anticancer therapies
* Documented or symptomatic brain or leptomeningeal metastasis
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency
* Previous treatment with monoclonal antibody therapy, other signal transduction inhibitors or epidermal growth factor receptor (EGFR) targeting therapy
* Evidence of previous other malignancy within the last 5 years
* Intake of any investigational medication within 30 days before trial entry
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Gao, Principal Investigator — Radiotherapy Department, Cancer Institute & Hospital, Chinese Academy of Medical Science, Beijing, China; Junliang Cai, Study Director — Merck Serono (Beijing) Pharmaceutical R&D Co., Ltd., an Affiliate of Merck KGaA, Darmstadt, Germany; Guozhen Xu, Principal Investigator — Radiotherapy Department, Cancer Institute & Hospital, Chinese Academy of Medical Science, Beijing, China
Locations (8):
- China (8):
  - Fujian Provincial Tumor Hospital, Fuzhou, Fujian
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhejiang Provincial Cancer Hospital, Hangzhou
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 70 participants were screened, out of which 4 participants were not treated and 66 participants received the study treatment.
Groups:
- Cetuximab: Participants received cetuximab 400 milligram/square meter (mg/m^2) intravenous (IV) infusion over 120 minutes for 1 week, subsequently followed by 250 mg/m^2 IV infusion over 60 minutes, from week 2 to 7 along with concomitant boost radiotherapy (RT): 72.0 Gray (Gy) total for 42 fractions in 6 weeks, initially, once-daily fractions: 32.4 Gy in 18 fractions of 1.8 Gy for 3.6 weeks (5 fractions/week), followed by twice-daily fractions 39.6 Gy in 24 fractions for 2.4 weeks: morning dose 1.8 Gy/fraction for a total of 12 fractions 5 fractions/week; evening dose 1.5 Gy/fraction for a total of 12 fractions 5 fractions/week. Doses were separated by at least a 6-hour interval.
Period: Overall Study
Arm/Group | Cetuximab
Started | 66
Completed | 0
Not Completed | 66
Not completed — Death | 14
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Progressive Disease (PD) | 18
Not completed — Symptomatic Deterioration | 1
Not completed — Another Anti-cancer Drug Received | 1
Not completed — Another Tumor Discovered | 1
Not completed — Ongoing | 29

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (9.5)
Age, Customized [Number; unit: participants]
  <65 years | 52
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR)
Description: Best overall (objective) response was defined as the occurrence of complete response (CR) or partial response (PR) based on the investigator's assessment according to modified World Health Organization (WHO) criteria confirmed at a repeat assessment performed no less than 28 days after the criteria for response were first met. CR was defined as disappearance of all index lesions. PR was defined as a 50% or more decrease in the sum of the products of diameters (SOPD) of index lesions compared to the baseline SOPD, with no evidence of PD.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 3 months following the 8 weeks after the end of RT visit until the end of trial (EOT) visit
Population: Intention-to-treat (ITT) population included all participants who received at least one dose of the investigational medicinal product (IMP) cetuximab or RT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 66
percentage of participants | 68.2 [55.6 to 79.1]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the duration (in months) from first administration of trial treatment to first observation of PD (radiological or clinical, if radiological PD is not available), or death due to any cause. The PFS time of participants without observation of PD but death occurring after two or more missed consecutive tumor assessments (i.e. two-fold scheduled time interval of two consecutive tumor assessments) was censored on the date of last tumor assessment or first administration of trial treatment (whichever was later).
Time Frame: Baseline up to disease progression or withdrawal or 12 weeks after the last radiotherapy of the last participant
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or RT.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 66
months | 9.4 [7.7 to 11.2]

ADVERSE EVENTS:
Time Frame: Up to Day 60 after last trial treatment administration and before EOT
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP, regardless of causal relationship and even if no IMP has been administered.
Groups:
- Cetuximab: Treatment Emergent Phase: Participants received cetuximab 400 milligram/square meter (mg/m^2) intravenous (IV) infusion over 120 minutes for 1 week, subsequently followed by 250 mg/m^2 IV infusion over 60 minutes, from week 2 to 7 along with concomitant boost radiotherapy: 72.0 Gray (Gy) total for 42 fractions in 6 weeks, initially, once-daily fractions: 32.4 Gy in 18 fractions of 1.8 Gy for 3.6 weeks (5 fractions/week), followed by twice-daily fractions 39.6 Gy in 24 fractions for 2.4 weeks: morning dose 1.8 Gy/fraction for a total of 12 fractions 5 fractions/week; evening dose 1.5 Gy/fraction for a total of 12 fractions 5 fractions/week. Doses were separated by at least a 6-hour interval. Treatment emergent phase, i.e. treatment-emergent adverse events (TEAEs, adverse events which occur or worsen on the first dosing day of trial treatment and until 60 days after the last trial treatment administration (cetuximab or radiotherapy).
- Cetuximab: Late Phase: Participants received cetuximab 400 milligram/square meter (mg/m^2) intravenous (IV) infusion over 120 minutes for 1 week, subsequently followed by 250 mg/m^2 IV infusion over 60 minutes, from week 2 to 7 along with concomitant boost radiotherapy: 72.0 Gray (Gy) total for 42 fractions in 6 weeks, initially, once-daily fractions: 32.4 Gy in 18 fractions of 1.8 Gy for 3.6 weeks (5 fractions/week), followed by twice-daily fractions 39.6 Gy in 24 fractions for 2.4 weeks: morning dose 1.8 Gy/fraction for a total of 12 fractions 5 fractions/week; evening dose 1.5 Gy/fraction for a total of 12 fractions 5 fractions/week. Doses were separated by at least a 6-hour interval. Late phase, i.e. adverse events which occur or worsen more than 60 days after the last trial treatment administration (cetuximab or radiotherapy), and before end of trial.
Arm/Group | Cetuximab: Treatment Emergent Phase | Cetuximab: Late Phase
Serious Adverse Events (participants affected / at risk) | 5/66 | 14/62
Other Adverse Events (participants affected / at risk) | 64/66 | 20/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab: Treatment Emergent Phase (N=66) | Cetuximab: Late Phase (N=62)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Localized edema (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Lung infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Esophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab: Treatment Emergent Phase (N=66) | Cetuximab: Late Phase (N=62)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 15 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Salivary gland pain (Gastrointestinal disorders) | 1 | 0
Tongue exfoliation (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
Infusion related reaction (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 52 | 0
Pyrexia (General disorders) | 14 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Furuncle (Infections and infestations) | 2 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Rubella (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 0
Radiation myelopathy (Injury, poisoning and procedural complications) | 0 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 9 | 0
Alanine aminotransferase increased (Investigations) | 5 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 34 | 11
Weight increased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 10 | 2
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 9 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Genital pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 11 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 13 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin chapped (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All submissions by the PI for publication require the written permission from the sponsor. The PI commits to forward to the sponsor all documents intended for publication which contains data or results generated in connection with the study. Documents must be available at least 60 days before the planned submission date to allow for review. Any publication should follow the policy in the protocol. The PI shall not publish results derived from the study until the study has been reported in full.